CLINICAL TRIAL: NCT05828160
Title: Development and Validation of the Italian Version of Modified Barthel Index and of the Motricity Index Scales
Brief Title: Italian Version of the Motricity Index
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Sponsor
Other Study IDs: mBI - MI - Part A
Record Dates: First submitted 2023-02-03; First posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-01

CONDITIONS: Cross-Cultural Comparison; Validation Study; Reliability and Validity; Disability Physical

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to develop and validate the Italian version of the Motricity Index (MI-Italian), through the following steps:

* translation of the MI into Italian, by using the forward-backward translation approach, to produce a pre-final MI-Italian
* pre-pilot testing of the pre-final MI-Italian in a sample of ten health professionals (physicians and physiotherapists), who will be asked to judge the clarity of each item of the MI, including scoring instructions, to produce a final MI-Italian
* evaluation of the metric properties (internal consistency, inter- and intra-rater reliability, validity and responsiveness) of the final MI-Italian in a sample of subjects admitted to the Don Gnocchi Foundation in Florence for rehabilitation after stroke.

DETAILED DESCRIPTION:
The Motricity Index (MI), developed by Demeurisse et al. in 1980, is an ordinal method for measuring motor impairment in post-stroke hemiparesis, focusing on muscle strength of proximal and distal muscle groups of upper and lower extremity. Since its introduction, it has been widely used. However, despite unofficial versions circulating in clinical settings, there is currently no validated Italian version of the scale. This study aims to develop this version and to evaluate its metric properties in a sample of subjects who had a stroke.

A pre-final MI-Italian will be produced following established international guidelines (forward-backward translation, each step involving two different translators). This version will be tested in a group of health professionals (physicians and physiotherapists) who will be asked to judge the clarity of each item of the scale, including scoring instructions, using a dichotomous response (clear/unclear). Items that are judged unclear by more than 20 percent of the professionals will be revised by the multidisciplinary translation team to produce the final MI-Italian.

The final MI-Italian will then be administered to a sample of at least 100 subjects with stroke to assess its metric properties. Participants will be enrolled among patients admitted to the Don Gnocchi Foundation in Florence for stroke rehabilitation. To assess reliability, upon admission each patient will be independently assessed using the MI-Italian by two examiners, drawn at random from a group of ten physiotherapists. One of the two raters will administer the scale twice on consecutive days. Other evaluators will administer other clinical scales (Fugl-Meyer assessment, FMA; modified Barthel index, mBI; modified Rankin scale, mRS) to assess the validity of the MI-Italian. All raters will be blinded to all other assessments and to their previous assessment, if any. All the scales will be administered again at discharge, when participants will also be asked to indicate the perceived change since admission in their ability to move and use the paretic limbs. For the latter, a 7-points Global Rating of Perceived Change (GRPC) Lickert scale will be used.

The Cronbach's alpha will be used to estimate the internal consistency of the scale. To assess intra-rater and inter-rater reliability, the Intraclass Correlation Coefficient (ICC1,1), Standard Error of the Measurement (SEM) and Minimal Detectable Change with 95% Confidence (MDC95) will be computed. Criterion and construct validity will be assessed by computing the association between the MI-Italian and the FMA, the mBI and the mRS, at both admission and discharge. For responsiveness, the following indices will be calculated: 1) Guyatt Responsiveness Index (GRI); 2) Standardized Response Mean (SMR), both in the whole sample and in subgroups of participants with different outcome (improved, unchanged, worsened) based on the GPRC; 3) Minimal Clinically Important Difference (MCID). The latter will be derived using the ROC curve approach, using the patient's perceived change in his/her ability to move and use the paretic limbs as an anchor.

ELIGIBILITY:
The study is divided in two phases: A) pilot-testing of the pre-final MI-Italian, and B) verification of the metric properties (reliability, validity and responsiveness) of the final MI-Italian.

A) Pilot-test of the pre-final MI-Italian (verification of clarity of all items)

Inclusion criteria:

* being a physician or a physiotherapist with at least three years of experience in the functional assessment of subjects with stroke
* willingness to participate in the study

Exclusion criteria: none.

B) Study on the metric properties of the final MI-Italian

Participants (subjects who had a stroke): all subject consecutively admitted to the Don Gnocchi Foundation of Florence for rehabilitation after stroke (until the expected sample size is completed) who meet the following criteria.

Inclusion:

* age 18 years or older
* stroke outcomes such that they impact the person's ability to independently perform various basic activities of daily living
* willingness to participate in the study, with informed consent signed (by the support administrator/legal guardian, if necessary)

Exclusion:

* severe visual and/or auditory impairment that cannot be corrected
* cognitive impairment defined by a Mini Mental State Examination (MMSE) score <21;
* severe language impairment such that comprehension and performance of the task is prevented
* presence of signs of clinical instability, defined by a score greater than zero on the Clinical Instability Scale Raters: ten physiotherapists with at least three years of experience in the evaluation and treatment of subjects with stroke outcomes. Pairs of raters, equal in number to the number of patients enrolled, will be randomly drawn from this group, and each pair will be randomly assigned to a patient to be administered the MI-Italian Other examiners, also randomly drawn from the list of ten raters, will administer other clinical scales to participants to assess the validity of the MI-Italian.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A) In the pilot-testing, the pre-final MI-Italian will be tested for clarity on a sample of 10 health professionals (physicians and physiotherapists) working in stroke rehabilitation.
  B) The metric properties of the final MI-italian will be tested on a sample of at least 100 patients who had a stroke. Considering a possible dropout rate of 15 percent, 115 subjects are expected to be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Estimated)
Dates: Start 2023-05-15 (Estimated); Primary Completion 2023-12-15 (Estimated); Study Completion 2024-02-15 (Estimated)

PRIMARY OUTCOMES:
Internal Consistency - Baseline assessment | Assessment at admission (T0),
  Cronbach's alpha
Internal Consistency - Discharge assessment | Discharge (T1) assessment. Time of discharge will vary among participants, so a definite time point cannot be stated. On average, discharge is expected after 30 days from admission.
  Cronbach's alpha
Intra-rater reliability | Test and Retest assessments, conducted 1-3 days apart.
  One-way random-effects model sIngle measures Intraclass Correlation Coefficient (ICC1,1)
Inter-rater reliability | Admission assessment conducted independently by two raters 30-60 minutes apart.
  One-way random-effects model sIngle measures Intraclass Correlation Coefficient (ICC1,1)
Intra-rater reliability (error of measurement) | Test and Retest assessments, conducted 1-3 days apart.
  Standard Error of the Measurements (SEM), computed as the standard deviation of the two measures collected by the same rater, multiplied by the square root of 1 minus ICC.
Inter-rater reliability (error of measurement) | Admission assessment conducted independently by two raters 30-60 minutes apart.
  Standard Error of the Measurements (SEM), computed as the standard deviation of the measures collected by two independent raters, multiplied by the square root of 1 minus ICC.
Intra-rater reliability (Minimal Detectable Change) | Test and Retest assessments, conducted 1-3 days apart.
  Minimal Detectable Change at the 95 % confidence level (MDC 95), computed as the SEM multiplied by 1,96 multiplied by the square root of 2.
Inter-rater reliability (Minimal Detectable Change) | Admission assessment conducted independently by two raters 30-60 minutes apart.
  Minimal Detectable Change at the 95 % confidence level (MDC 95), computed as the SEM multiplied by 1,96 multiplied by the square root of 2.
Criterion Validity - Association with reference standard at admission. | Admission assessment (T0).
  Estimation of the correlation between the MI-Italian and Motricity subsection of the Fugl Meyer Assessment (FMA) scale, separately for upper limb and lower limb.
Criterion Validity - Association with reference standard at discharge | Discharge (T1) assessment. Time of discharge will vary among participants, so a definite time point cannot be stated. On average, discharge is expected after 30 days from admission.
  Estimation of the correlation between the MI-Italian and Motricity subsection of the Fugl Meyer Assessment (FMA) scale, separately for upper limb and lower limb.
Construct validity (Hypothesis testing) - Association with function at admission | Admission assessment (T0).
  Estimation of the correlation between the total scores of the MI-Italian and the modified Barthel Index (mBI).
Construct validity (Hypothesis testing) - Association with function at discharge. | Discharge (T1) assessment. Time of discharge will vary among participants, so a definite time point cannot be stated. On average, discharge is expected after 30 days from admission.
  Estimation of the correlation between the total scores of the MI-Italian and the modified Barthel Index (mBI).
Responsiveness (change of MI-Italian scores from admission to discharge) - Standardized Response Mean (SRM). | Admission (T0) and Discharge (T1) assessment. Time of discharge will vary among participants, so a definite time point cannot be stated. On average, discharge is expected after 30 days from admission.
  For each subject, the change score at the MI-Italian will be calculated as the difference between T1 and T0 assessment. The SRM will be calculated as the ratio of observed change and the standard deviation reflecting the variability of the change scores, both in the whole sample and separately in groups with different outcome based on the Global Rating of Perceived Change (GRPC).
Responsiveness (change of MI-Italian scores from admission to discharge) - Guyatt Responsiveness Index (GRI) | Admission (T0) and Discharge (T1) assessment. Time of discharge will vary among participants, so a definite time point cannot be stated. On average, discharge is expected after 30 days from admission.
  For each subject, the change score at the MI-Italian will be calculated as the difference between T1 and T0 assessment. The GRI will be calculated as the ratio of the mean change score difference between improved and stable patients and the standard deviation of the individual change scores in stable patients. Improved and stable patients will be detected based on the GRPC.
Responsiveness (change of MI-Italian scores from admission to discharge) - Minimal Clinically Important Difference (MCID). | Admission (T0) and Discharge (T1) assessment. Time of discharge will vary among participants, so a definite time point cannot be stated. On average, discharge is expected after 30 days from admission.
  For each subject, the change score at the MI-Italian will be calculated as the difference between T1 and T0 assessment. The Receiving Operator Characteristic (ROC) curve approach will be used to estimate the minimal change score associated with clinically important change (i.e., the MCID), using the GRPC as an anchor.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Beaton DE, Bombardier C, Guillemin F, Ferraz MB. Guidelines for the process of cross-cultural adaptation of self-report measures. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3186-91. doi: 10.1097/00007632-200012150-00014. No abstract available. PMID 11124735
- [Background] Bertrand AM, Fournier K, Wick Brasey MG, Kaiser ML, Frischknecht R, Diserens K. Reliability of maximal grip strength measurements and grip strength recovery following a stroke. J Hand Ther. 2015 Oct-Dec;28(4):356-62; quiz 363. doi: 10.1016/j.jht.2015.04.004. Epub 2015 May 9. PMID 26206167
- [Background] Cameron D, Bohannon RW. Criterion validity of lower extremity Motricity Index scores. Clin Rehabil. 2000 Apr;14(2):208-11. doi: 10.1191/026921500675786655. PMID 10763800
- [Background] Collin C, Wade D. Assessing motor impairment after stroke: a pilot reliability study. J Neurol Neurosurg Psychiatry. 1990 Jul;53(7):576-9. doi: 10.1136/jnnp.53.7.576. PMID 2391521
- [Background] Demeurisse G, Demol O, Robaye E. Motor evaluation in vascular hemiplegia. Eur Neurol. 1980;19(6):382-9. doi: 10.1159/000115178. PMID 7439211
- [Background] Fayazi M, Dehkordi SN, Dadgoo M, Salehi M. Test-retest reliability of Motricity Index strength assessments for lower extremity in post stroke hemiparesis. Med J Islam Repub Iran. 2012 Feb;26(1):27-30. PMID 23483112
- [Background] Gor-Garcia-Fogeda MD, Molina-Rueda F, Cuesta-Gomez A, Carratala-Tejada M, Alguacil-Diego IM, Miangolarra-Page JC. Scales to assess gross motor function in stroke patients: a systematic review. Arch Phys Med Rehabil. 2014 Jun;95(6):1174-83. doi: 10.1016/j.apmr.2014.02.013. Epub 2014 Feb 28. PMID 24582618
- [Background] Jacob-Lloyd HA, Dunn OM, Brain ND, Lamb SE. Effective Measurement of the Functional Progress of Stroke Clients. British Journal of Occupational Therapy. 2005;68(6):253-259. doi:10.1177/030802260506800603
- [Background] Lin C, Arevalo YA, Harvey RL, Prabhakaran S, Martin KD. The minimal clinically important difference of the motricity index score. Top Stroke Rehabil. 2023 Apr;30(3):298-303. doi: 10.1080/10749357.2022.2031532. Epub 2022 Jan 30. PMID 35094664
- [Background] Sousa VD, Rojjanasrirat W. Translation, adaptation and validation of instruments or scales for use in cross-cultural health care research: a clear and user-friendly guideline. J Eval Clin Pract. 2011 Apr;17(2):268-74. doi: 10.1111/j.1365-2753.2010.01434.x. Epub 2010 Sep 28. PMID 20874835
- [Background] Sunderland A, Tinson D, Bradley L, Hewer RL. Arm function after stroke. An evaluation of grip strength as a measure of recovery and a prognostic indicator. J Neurol Neurosurg Psychiatry. 1989 Nov;52(11):1267-72. doi: 10.1136/jnnp.52.11.1267. PMID 2592969
- [Background] Vos-Vromans DC, de Bie RA, Erdmann PG, van Meeteren NL. The responsiveness of the ten-meter walking test and other measures in patients with hemiparesis in the acute phase. Physiother Theory Pract. 2005 Jul-Sep;21(3):173-80. doi: 10.1080/09593980500212920. PMID 16389698
- [Background] Wade DT, Hewer RL. Functional abilities after stroke: measurement, natural history and prognosis. J Neurol Neurosurg Psychiatry. 1987 Feb;50(2):177-82. doi: 10.1136/jnnp.50.2.177. PMID 3572432